CLINICAL TRIAL: NCT04741100
Title: Evaluation of Innovative Combinatorial stratégies of Anti-latency and Anti-immune Activation Drugs Targeting HIV Reservoir
Acronym: ERAVIR
Status: Withdrawn | Type: Observational
Why Stopped: No patients Enrolled
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 04
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ex-vivo analysis — Ex-vivo analysis

SUMMARY:
Several barriers prevent the remission of HIV infection: low level viremia, HIV latency in the genome of host infected immune cells and persistent immune activation. Targeting immune activation and viral latency, represent the two intimately intricate goals to be envisaged for purging the reservoir, in the perspective of HIV cure. There is an urgent to develop and to test drugs targeting HIV latency, HIV residual replication and immune activation, alone or in synergistic combinations.

We propose in this study to test agents with a potential effect on HIV latency by combining classical agents and newly discovered agents.

The Pitié-Salpêtrière virology group has identified some new diaminopiperidine based compounds that have some antilatency properties through an activation of transcription. Compounds of this new class will be tested in combination with classical agents (HDAC inhibitors, HMT inhibitors, inducers of P-TEFb release, PKC agonists, DNMT inhibitors) and less toxic compounds from classical categories for which Carine Van Lint (University of Brussels) has obtained preliminary HIV reactivation data.

All the experimentations will be conducted in J-Lat cells and in ex- vivo CD4 cells sampled in patients from the Pitié-Salpêtrière HIV cohort.

DETAILED DESCRIPTION:
Despite its major benefits, cART implies mandatory lifespan treatment, toxicity, high costs and the inability to restore full-health, thus urging the need to find a cure strategy and to revisit our approach to HIV therapy.

HIV eradication is currently not achievable with standard cART due to the persistence of HIV reservoir maintained through low-level viremia, immune activation despite plasma viral suppression and HIV latency.

The possibility to achieve HIV eradication has been limited, at least in part, by the existence of latently infected cellular reservoirs. The major known cellular reservoir is established in quiescent memory CD4+ T cells, providing an extremely long-lived set of cells in which the virus can remain transcriptionally silen. Reactivation of latent viruses followed by the killing of the infected cells has been proposed as a possible strategy (''shock and kill'') to purge the latent reservoir. None of them have been currently really successful. Innovative strategies to target HIV reservoir are needed. In parallel to clinical interventions, there is a need to screen in vitro and ex vivo the best anti-latency and anti-immune activation candidates, thus defining the optimal strategy targeting the reservoir.

Research on the control of HIV latency and potential reactivation have been hindered by the small numbers of latently infected cells in vivo and the absence of known phenotypic markers to distinguish those cells from uninfected cells. In this setting, cell-line models of latency have been very useful due to their genetic and experimental tractability. Major conceptual leaps have been facilitated by the use of latently infected T cell lines, including the ability to conduct genetic screens. On the other hand, latently infected cell lines are limited by their cycling nature and inherent mutations in growth controls, and the clonal nature of the virus integration sites. Such transformed cell lines lack the ability to differentiate and naturally oscillate between phases of quiescence and active proliferation in response to biological signals. Because of these limitations, several laboratories have recently developed primary cellular models of HIV-1 latency that capitalize on specific aspects of the T cell reservoir, found in vivo. These newer models allow easily and rapidly to study proposed virological and cellular mechanisms of latency and to evaluate novel small molecule compounds for induction of viral reactivation.

One particular complex issue is the diversity of latency models and the many differences among them. Disparities relate to: the T-cell subsets represented; the cellular signaling pathways capable of driving viral reactivation; and the genetic composition of the viruses employed, ranging from wild-type to functional deletion of multiple genes. Additional differences reside in the experimental approaches taken to establish latent infection in these primary cell models, which involve either infection of activated cycling cells later allowed to return to a resting state, or direct infection of quiescent cells. Because of such system variables, screening efforts in specific cell models with identified drug candidates for ''anti-latency'' therapy often fail to reactivate HIV uniformly across the different models. Therefore, the activity of a drug candidate, varies from one cellular model, to another one or in cells from infected patients, tested ex-vivo. The current situation in this research field represents a critical knowledge gap that is adversely affecting our ability to identify promising treatment compounds and their associated molecular mechanisms and is hindering the advancement of drug testing into relevant animal models and ultimately, human clinical trials.

In a recent study, induction of viral reactivation across several cell models was assessed using a selected common panel of stimuli known to function by distinct and defined mechanisms of action. The panel included 13 treatments that modulate T cell processes such as T-cell receptor engagement, protein kinase C (PKC) activation, calcium influx, cytokine signaling, histone deacetylation, and release of P-TEFb from the HEXIM/7SK RNP complex. This last study was designed to answer the following questions: 1) are certain models of latency biased towards or against particular cell signaling pathways? 2) can stimuli that work uniformly in multiple models be identified? 3) can a central uniting theme or a single signaling pathway be responsible for control of viral latency? and 4) can a model or limited group of models predict experimental drug activity in authentic latently infected cells from patients? The results indicate that no single in vitro cell model alone is able to capture accurately the ex vivo response characteristics of latently infected T cells from patients. Most cell models demonstrated that sensitivity to HIV reactivation was skewed towards or against specific drug classes. Protein kinase C agonists and PHA reactivated latent HIV uniformly across models, although in most other drug classes did not.

From these observations, it is obvious that single agents will not be enough potent to induce an efficient stimulation of HIV transcription and latency disruption.

We propose in the Eravir study to test several agents in combinations including classical agents and new classes of agents recently discovered in our institutions in their capacity to reactivate HIV.

All experimentations will be conducted in J-Lat cells and in ex vivo CD4 cells sampled in HIV patients with a fully suppressed viremia on antiretroviral treatment.

The team of Pitié-Salpêtrière has identified some new compounds diaminopiperidine based that have some properties that could disturb latency of HIV allowing an activation of transcription. Compounds of this family will be tested in combination with classical agents such as HDAC inhibitors, HMT inhibitors, inducers of P-TEFb release, PKC agonists, DNMT inhibitors and also with compounds from these categories but less toxic for which Carine Van Lint's lab (University of Brussels) has obtained preliminary HIV reactivation data.

All the tests will be conducted in J-Lat cells and in ex vivo CD4 cells sampled in patients of Pitié-salpêtrière Hospital (Paris) and of Saint-Pierre Hospital (Bruxells).

Also frozen viable PBMC-samples will be dispatched from Belgium and France to the Spanish partner in order to test immune-activation and inflammation parameters.

The research question will evaluate whether these above mentioned combination are capable to reactivate HIV from cellular models and ex vivo in patient cells.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* CD4+ count nadir ≥ 200 cells/mm3
* At least 4 years of suppressive ART, i.e. HIV plasma viral load (RNA) ≤ 50 copies/ml without any interruption (less than one month cumulative);1 blip/year allowed at values of maximum 1000 cp/ml
* CD4+ count ≥ 500 cells/mm3 in the 6 months prior to inclusion
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Active HBV and/or HCV co-infection
* Pregnancy or breast-feeding woman
* Previous immunotherapy (e.g. IL-2, IL-7) within the past year
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* History of autoimmune disease, such as systemic lupus erythematosis (SLE) or Hashimoto's thyroiditis
* Active drug or alcohol use or dependence that, in the opinion of the center investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients HIV infected on suppressive cART
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome Measure | 18 months
  Measure the new anti-latency drugs to assess ex vivo the synergistic effects of from different families in different cells

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Pitie-Salpetriere Hospital